CLINICAL TRIAL: NCT00544141
Title: Clinical Evaluation of the Care On Line Thermometer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medisim Ltd (Industry)
Other Study IDs: 26-115-44
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Temperature measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical study is to evaluate the performance of the COL thermometer by comparing its measurement to equilibrium measurement and to make a final tuning of the thermometer algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-18 years old) in the pediatric or emergency department, with or without fever.
* An informed consent was signed by the patient's guardian.

Exclusion Criteria:

* The medical staff decides that participating will damage patient recovery.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children (1-18 years old) in the pediatric or emergency department, with or without fever.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Yehezkel Waisman, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel